CLINICAL TRIAL: NCT03726294
Title: A Phase 1, Open-label, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Efficacy of NBM-BMX in Subjects With Advanced Solid Tumors
Brief Title: A Safety and Pharmacokinetic Study of NBM-BMX Administered Orally to Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NatureWise Biotech & Medicals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBM-BMX-001
Record Dates: First submitted 2018-10-26; First posted 2018-10-31 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NBM-BMX (Experimental)
  Interventions: Drug: NBM-BMX softgel capsules

INTERVENTIONS:
Drug: NBM-BMX softgel capsules — Patients will initially receive NBM-BMX orally once a day at 100 mg per day.

SUMMARY:
NBM-BMX is a new small molecule chemical entity being developed as a potential anti-cancer therapeutic by NatureWise. NBM-BMX is a histone deacetylase (HDAC) inhibitor and has been shown to be particularly active against HDAC8. The objectives of this study are to determine the safety profile of NBM-BMX, including identification of dose limiting toxicity (DLT) and maximum tolerated dose (MTD), and to determine the Recommended Phase 2 Dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced, non-resectable, and/or metastatic solid tumor refractory to standard of care therapy, or for whom no standard of care therapy is available, or who were not amenable to established forms of treatment.
2. Solid tumors must have measurable or evaluable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
3. Female or male at 18 years of age or older.
4. ECOG performance status 0 to 2.
5. Recovered from prior treatment-related toxicity to at least grade 1 with exception of grade 2 alopecia or other grade 2 toxicity with prior approval of the Medical Monitor.
6. Adequate organ function as defined by the following criteria:

   * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤3 x upper limit of normal (ULN), or AST and ALT ≤5 x ULN if liver function abnormalities are due to underlying malignancy
   * Total serum bilirubin ≤1.5 x ULN (except for subjects with documented Gilbert's syndrome)
   * Absolute neutrophil count (ANC) ≥ 1500/μL
   * Platelets ≥ 90,000/μL
   * Hemoglobin ≥ 9.0 g/dL
   * Serum creatinine ≤1.5 x ULN or creatinine clearance of ≥ 60 mL/min
7. Signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment.
8. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the trial:

1. Major surgery or radiation therapy within 28 days of starting study treatment.
2. Systemic anti-cancer therapy within 28 days or 5 half-lives (whichever is shorter) of starting study treatment.
3. Prior high-dose chemotherapy requiring hematopoietic stem cell rescue.
4. Current treatment on another clinical trial.
5. Spinal cord compression, carcinomatous meningitis, or leptomeningeal disease unless appropriately treated and neurologically stable for at least 4 weeks.
6. Any of the following within the 12 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack; within 6 months prior to starting study treatment for pulmonary embolus. However, upon agreement between the investigator and sponsor, the 6 month post-event-free period for a subject with a pulmonary embolus can be waived if due to advanced cancer. Appropriate treatment with anticoagulants is permitted.
7. NYHA Class III or IV heart failure and known history of QTc prolongation or Torsade de Pointes.
8. Use of medications known to significantly prolong the QTc interval (e.g., antiarrhythmic and psychotropic medications).
9. Hypertension that cannot be controlled by medications.
10. Current treatment with therapeutic doses of warfarin (low dose warfarin up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed).
11. Known human immunodeficiency virus (HIV)-positive and is receiving antiretroviral therapy. Subjects with known HIV infection and on a stable dose of HIV suppressive medication may be eligible if considered to be at low risk for AIDS-related outcomes following discussion with the medical monitor.
12. Known hepatitis B virus (HBV) or hepatitis C virus (HCV) with evidence of chronic active disease or receiving/requiring antiviral therapy.
13. History of receiving organ transplantation or immune disorders that require continuous immunosuppressant agent therapy.
14. Pregnancy or breastfeeding. Female subjects must be surgically sterile or be postmenopausal, or must agree to the use of effective contraception during the period of therapy. All female subjects with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
15. Other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that would impart, in the judgment of the investigator and/or sponsor, excess risk associated with study participation or study drug administration, which would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) of NBM-BMX [Safety and Tolerability] | up to 28 days
  Toxicities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0
Maximum tolerated dose (MTD) of NBM-BMX [Safety and Tolerability] | up to 28 days
  The MTD will be defined as the dose level at which at most one of six patients experiences a DLT after 28 days of treatment have occurred, with the next higher dose having at least 2/3 or 2/6 patients experiencing a DLT.

SECONDARY OUTCOMES:
Preliminary assessment of anti-tumor activity by Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) [Efficacy] | at least 8 weeks
AUC(0-last) of NBM-BMX [Pharmacokinetics] | Day 1, 8 and 15 for Cycle 1 only (each cycle is 28 days)
  AUC(0-last): area under the plasma concentration versus time curve to the time of the last measurable concentration
Cmax of NBM-BMX [Pharmacokinetics] | Day 1, 8 and 15 for Cycle 1 only (each cycle is 28 days)
  Cmax: maximum plasma concentration
Tmax of NBM-BMX [Pharmacokinetics] | Day 1, 8 and 15 for Cycle 1 only (each cycle is 28 days)
  Tmax: time to maximum plasma concentration
T(1/2) of NBM-BMX [Pharmacokinetics] | Day 1 and 15 for Cycle 1 only (each cycle is 28 days)
  T(1/2): terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Anthony W. Tolcher, M.D., Principal Investigator — NEXT Oncology
Locations (1):
- NEXT Oncology, San Antonio, Texas, United States